CLINICAL TRIAL: NCT05773040
Title: A Phase 1 Study of JV-213 Autologous CD79b-targeting Chimeric Antigen Receptor T-cell Therapy in Adults With Relapsed or Refractory B-cell Lymphomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0938; NCI-2023-02055 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-03-01; First posted 2023-03-17 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Lymphomas; B-cell Lymphomas
Keywords: B-cell lymphoma, CD79b, CAR T cell therapy
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell | interventions — Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 (dose escalation) (Experimental): Part 1, the dose of JV-213 participants receive will depend on when you join this study. Up to 3 dose levels of JV-213 will be tested. About 3-6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level of JV-213. Each new group will receive a higher dose of JV-213 than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of JV-213 is found.
  Interventions: Drug: JV-213; Procedure: Leukapheresis
- Part 2 (dose expansion) (Experimental): Participants will receive JV-213 at the recommended dose that was found in Part 1.
  Interventions: Drug: JV-213; Procedure: Leukapheresis

INTERVENTIONS:
Drug: JV-213 — Given by (IV) vein
Procedure: Leukapheresis — Given by IV (vein)

SUMMARY:
To find the highest tolerable dose of JV-213 (a type of autologous CAR T cell therapy) that can be given to patients who have B-cell lymphoma that is relapsed or refractory.

DETAILED DESCRIPTION:
Primary Objectives:

--The primary objective is to determine the safety and identify the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of JV-213 in patients with r/r B-cell lymphomas.

Hypothesis: JV-213 will be safe, well-tolerated, and effective in patients with r/r B-cell lymphomas.

Secondary Objectives:

--The secondary objective is to determine the efficacy in adults with r/r LBCL and FL grade 3B treated at the MTD or RP2D of JV-213. Although the clinical benefit of JV-213 has not yet been established, the intent of offering this treatment is to provide a possible therapeutic benefit, and thus the patient will be carefully monitored for tumor response and symptom relief in addition to safety and tolerability. Secondary endpoints include overall response rate (ORR; including CR + PR) and CR rate as defined by the Lugano Classification response criteria for malignant lymphoma,53 DOR, PFS, and OS.

Hypothesis: JV-213 will induce an ORR of at least 40% in adult subjects with r/r B-cell lymphomas.

Exploratory Objectives:

--The exploratory objectives are to assess the cellular kinetics and pharmacodynamic effects of JV-213 anti-CD79b CAR T-cell product and to evaluate biomarkers associated with response, resistance, and toxicity after administration of JV-213 in blood and tumor samples.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following inclusion criteria in order to be eligible for participation in this trial:

1. For the dose escalation cohort: Eligible patients will include those with r/r B-cell lymphoma including LBCL (DLBCL, HGBCL, LBCL transformed from indolent lymphoma, and PMBCL), FL, marginal zone lymphoma, and MCL after at least 2 prior systemic therapies and Burkitt lymphoma after at least 1 prior systemic therapy. For the dose expansion cohort: Patients with r/r LBCL (DLBCL, HGBCL, LBCL transformed from indolent lymphoma, and PMBCL) and FL grade 3B will be eligible
2. Received at least 2 prior lines of therapy, including anti-CD20 antibody and anthracycline therapy for LBCL, anti-CD20 antibody and alkylating agent or lenalidomide therapy for FL, anti-CD20 antibody and alkylating agent or lenalidomide or BTK inhibitor therapy for marginal zone lymphoma, and anti-CD20 antibody and alkylating agent or BTK inhibitor therapy for MCL. Patients with Burkitt lymphoma may be eligible after 1 line of prior therapy including anti-CD20 antibody and anthracycline therapy.
3. Patients who have received prior CD19 CAR cell therapy using FMC63 antibody for targeting CD19 are eligible and must be at least 6 weeks post CAR infusion and have <5% of peripheral blood T cells expressing the prior CAR by flow cytometry assessment.
4. ≥18 years of age
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
6. At least one measurable lesion per the Lugano 2014 Classification53
7. At least two weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic anti-cancer therapy prior to leukapheresis. For patients treated with monoclonal antibody-based therapies, at least 4 weeks must have elapsed prior to leukapheresis.
8. Toxicities due to prior therapy must be stable and recovered to ≤grade 1 (except for clinically non-significant toxicities such as alopecia)
9. Absolute neutrophil count of ≥1.0×10^9/L
10. Absolute lymphocyte count of ≥0.1×10^9/L
11. Platelet count of ≥75×10^9/L
12. Creatinine clearance (as estimated by Cockcroft Gault) ≥45 mL/min
13. Serum alanine transaminase (ALT) / aspartate transaminase (AST) ≤5 times the upper limit of normal (ULN)
14. Total bilirubin ≤2 mg/dL, except in patients with Gilbert's syndrome.
15. Cardiac ejection fraction ≥45% with no evidence of clinically significant pericardial effusion
16. Baseline oxygen saturation ≥92% on room air
17. Women of childbearing potential must have a negative serum or urine pregnancy test (women who have had hysterectomy and women who are over the age of 45 years and

Exclusion Criteria:

Patients will be excluded from participating in the trial if he/she has:

1. Active central nervous system (CNS) lymphoma including patients with detectable cerebrospinal fluid malignant cells or brain metastases. Patients with prior CNS lymphoma that has been effectively treated will be eligible if treatment was completed at least one year prior to enrolment and there is no evidence of disease on MRI with gadolinium contrast at the time of screening.
2. Any CAR cell therapy using non-FMC63 antibody.
3. History of Richter's transformation of chronic lymphocytic leukemia
4. Autologous stem cell transplantation within 6 weeks.
5. Allogeneic stem cell transplantation within 3 months or active graft versus host disease.
6. Active autoimmune disease (e.g. Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) requiring systemic immunosuppression/systemic disease modifying agents within the last 1 year or inflammatory disease (including graft versus host disease) requiring systemic immunosuppressive therapy. Physiological replacement of corticosteroids of up to 7.5 mg of prednisone or equivalent per day, and topical and inhaled corticosteroids are permitted.
7. History of any form of primary immunodeficiency that in the opinion of the investigator may affect efficacy of the CAR-T product.
8. History of any one of the following cardiovascular conditions within the past 6 months: Class III or IV heart failure as defined by the New York Heart Association, cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease.
9. History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) unless disease free for at least 2 years and treated with curative intent. Patients with a prior history of malignancy whose natural history or treatment (e.g. hormonal therapy) does not have the potential to interfere with either the safety or efficacy assessment of the investigational regimen in the opinion of the investigator may be included.
10. Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous antimicrobials for management. Simple urinary tract infection and uncomplicated bacterial pharyngitis or localized skin infections are permitted if responding to active treatment and after consultation with the Principal Investigator.
11. Known history of infection with HIV or hepatitis B (HBsAg positive) or hepatitis C virus (anti-HCV positive). A history of hepatitis B or hepatitis C is permitted if the viral load is undetectable per quantitative PCR and/or nucleic acid testing.
12. History or presence of CNS disorders such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement
13. Patients with cardiac atrial or cardiac ventricular lymphoma involvement
14. Requirement for urgent therapy due to tumor mass effect such as bowel obstruction or blood vessel compression
15. Any medical condition likely to interfere with assessment of safety or efficacy of study treatment
16. Live vaccine ≤6 weeks prior to planned start of conditioning regimen
17. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the conditioning chemotherapy on the fetus or infant.
18. Females of childbearing potential and males of child fathering potential who are not willing to practice two methods of birth control from the time of consent through 6 months after infusion of the study drug
19. In the investigator's judgment, the patient is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sattva Neelapu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-09-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT05773040/ICF_000.pdf